CLINICAL TRIAL: NCT03488056
Title: Effectiveness of the International Caries Classification and Management System (ICCMS) in Reducing the Incidence of Dental Caries in Children Attending to the CURUMIM Social Project, Sesc/São Paulo(SP)
Brief Title: Effectiveness of ICCMS in Reducing the Incidence of Dental Caries in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Serviço Social do Comércio - SESC (Unknown)
Responsible Party: Principal Investigator, Mariana Minatel Braga, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CURUMIM
Record Dates: First submitted 2018-03-20; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Dental Caries
Keywords: Dental Caries, ICCMS, Risk Assessment
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: The randomization was made by centers of the SESC (Social Service of the Commerce) of São Paulo state. Four centers will follow the ICCMS criteria and four other centers will follow criteria for diagnosis and treatment of SESC. The randomization will be stratified by sociodemographical conditions. The minimization will be used to equate preexisting oral health-related activities. According to allocated strategy, dentists in the center will guide their conduct with children attended to the CURUMIM project.
Who Masked: Participant, Outcomes Assessor
Masking Description: The division of the control and experimental groups was done by center and for neither group are revealed to the patient nor responsible for the type of intervention they are undergoing.
  After a certain time of the study, a blind investor will examine the children's centers and evaluate the outcome of the study. This researcher will not know which center is a control or experimental group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - ICCMS (Experimental): The dentists will perform clinical examination on children following the ICCMS sequence:
  The patient's caries risk assessment, Diagnosis of caries lesion and activity assessment Intraoral risk assessment, Decide on a personalized care plan for patient and clinical interventions.After asses all the factors and defining the patient's individual risk, the system presents a personalized treatment plan, indicating the appropriate home care instructions, clinical interventions and specific treatment for each caries lesion categories.
  The return intervals will be scheduled according to the risk: low risk (return of 1 year), moderate risk (6 months) and high risk (3 months)
  Interventions: Other: ICCMS
- Control - Standard care SESC (Active Comparator): The clinical sequence in this group will be:
  Caries Diagnosis Operative and non-operative treatments Indication of recall interval according to the dentist However, dentists will do that without a schematic guide to follow. They will do as they usually do in their practices.
  Interventions: Other: SESC standard care

INTERVENTIONS:
Other: ICCMS — The patient's caries risk assessment, Diagnosis of caries lesion and activity assessment
  -Intraoral risk assessment, Decide on a personalized care plan for patient and clinical interventions.
  After asses all the factors and defining the patient's individual risk, the system presents a personalized treatment plan, indicating the appropriate home care instructions, clinical interventions and specific treatment for each caries lesion categories.
  The treatment is divided into Non-Operative Care and Tooth-Preserving Operative Care (restorations with minimal intervention to preserve maximum dental structure).
  The return intervals will be scheduled according to the risk: low risk (return of 1 year), moderate risk (6 months) and high risk (3 months)
  Arms: Test - ICCMS
Other: SESC standard care — Standard care related to: Caries Diagnosis, operative and non-operative treatments, Indication of recall interval according to the dentist opinion
  Arms: Control - Standard care SESC

SUMMARY:
The aim of the present study is to evaluate the effectiveness of using the ICCMS (International Caries Classification And Management System)in reducing caries lesions incidence compared to a control group that use different criteria as a not systematic and standardized prevention strategy. The study will be performed among children attending to the social project of Social Service of Commerce (SESC), Sao Paulo. The sample will be composed of 460 children aging between 7 to 12 years old registered in CURUMIM Program from eight dental centers of SESC. A randomized controlled study with parallel group will be conducted. The centers will be randomized between the 2 strategies, defining 2 groups with 4 centers each. The experimental group that will follow the criteria defined by the ICCMS will evaluate clinical and behavioral variables, it will define: evaluation of the caries risk of the patient, evaluation of the intraoral risk, diagnosis of the caries lesion and its respective activity, plan decision individualized treatment for the patient and indication of recall interval according to the risk of caries. In the control group, children need will be solved according to rthe routinely dental practices in the center, but the determination of the child's general and intraoral risk of developing new caries lesions will not be performed nor the scheduling of specific recall intervals according to the risk.

ELIGIBILITY:
Inclusion Criteria:

* Children who participate in the CURUMIM Program
* Children whose parents sign the term of informed consent confirming their participation.

Exclusion Criteria:

* Children with cognitive impairment, motor impairment and feeding tube.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 460 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of caries | 2 years
  New cavitated caries lesions
Cost-effectiveness | 2 years
  Ratio between the difference in costs and in effects regarding the programs

SECONDARY OUTCOMES:
New initial caries lesions | 2 years
  New initial caries lesions
Qualitative measurement of difficulties and issues during the programs implementation | 2 years
  Health professional views about the program implementation (impact) collected periodically by a structured online report followed by an interview
Oral Health-Related Quality of Life (OHRQoL) | 2 years
  Difference in Oral Health-Related Quality of Life (OHRQoL) scores using the Brazilian validated version of Early Childhood Oral Health Impact Scale (ECOHIS) questionnaire (before and after treatment). Bigger the difference, bigger the impact of the program on children's OHRQoL

CONTACTS AND LOCATIONS:
Overall Officials: Mariana M Braga, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, Brazil